CLINICAL TRIAL: NCT01921088
Title: Real-Time Functional Magnetic Resonance Imaging Neurofeedback for Regulation of Psychophysiological Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Swiss National Science Foundation (Other); Korea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NF1_137023_A
Record Dates: First submitted 2013-08-02; First posted 2013-08-13 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Stress; Blood Pressure
Keywords: fMRI; Neurofeedback; Blood pressure; Psychophysiology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingent (Experimental): Contingent RT-fMRI-NF of brain activity in the target region of interest
  Interventions: Other: real-time functional magnetic resonance imaging neurofeedback (RT-fMRI-NF); Behavioral: Ambulatory Training
- Non-contingent (Sham Comparator): Sham RT-fMRI-NF of brain activity of previously recorded subject
  Interventions: Other: real-time functional magnetic resonance imaging neurofeedback (RT-fMRI-NF); Behavioral: Ambulatory Training

INTERVENTIONS:
Other: real-time functional magnetic resonance imaging neurofeedback (RT-fMRI-NF) — Subjects are provided with RT-fMRI-NF.
  Other Names: There are no specific branded names etc. associated with the intervention.
Behavioral: Ambulatory Training — Subjects are provided with an ambulatory training.

SUMMARY:
The purpose of this study is to determine the potential efficacy of real-time functional magnetic resonance imaging neurofeedback (RT- functional magnetic resonance imaging (fMRI) -NF) in regulating brain activity and psychophysiological functions.

DETAILED DESCRIPTION:
The overall goal of the outlined study is to establish a real-time functional magnetic resonance imaging neurofeedback (RT-fMRI-NF) protocol aiming at modulating brain activity and psychophysiological functions. About two weeks after the initial training session it will be estimated how stable training effects have been. The two weeks in between, subjects will receive ambulatory training of the strategies via a smartphone-based application.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient spoken and written knowledge of English
* Right-handedness
* Access to smartphone
* Availability to participate in the study

Exclusion Criteria:

* Color blindness
* Presence of cardiovascular disease
* Medication intake affecting cardiovascular function
* Medical MRI contraindication

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-08; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure | study day 1; study day 2 (2 weeks later); anticipated: follow-up (up to 1 year)
  assessed via oscillometry, expressed in mmHg
Blood oxygenation level dependent signal of the target brain region of interest | study day 1; study day 2 (2 weeks later); anticipated: follow-up (up to 1 year)
  blood oxygenation level dependent (BOLD) signal assessed via functional magnetic resonance imaging, expressed in relative BOLD signal intensity

SECONDARY OUTCOMES:
Feedback on adverse events during the scanner and ambulatory training | study day 1; study day 2 (2 weeks later); anticipated: follow-up (up to 1 year)
  number of subjects reporting an adverse event

OTHER OUTCOMES:
Psychobiological stress reactivity | study day 1; study day 2 (2 weeks later); anticipated: follow-up (up to 1 year)
  assessed via heart rate, cortisol
Psychological stress reactivity | study day 1; study day 2 (2 weeks later); anticipated: follow-up (up to 1 year)
  assessed via Multidimensional Mood State Questionnaire; Self-Assessment Manikin; Perceived Stress Scale
Functional connectivity | study day 1; study day 2 (2 weeks later); anticipated: follow-up (up to 1 year)
  connectivity of brain activity determined by fmri signal

CONTACTS AND LOCATIONS:
Overall Officials: Marion Tegethoff, PhD, Principal Investigator — University of Basel; Jong-Hwan Lee, PhD, Principal Investigator — Korea University; Gunther Meinlschmidt, PhD, Principal Investigator — University of Basel;Ruhr-University Bochum
Locations (1):
- Korea University, Seoul, South Korea

REFERENCES:
- [Derived] Meinlschmidt G, Lee JH, Stalujanis E, Belardi A, Oh M, Jung EK, Kim HC, Alfano J, Yoo SS, Tegethoff M. Smartphone-Based Psychotherapeutic Micro-Interventions to Improve Mood in a Real-World Setting. Front Psychol. 2016 Jul 28;7:1112. doi: 10.3389/fpsyg.2016.01112. eCollection 2016. PMID 27516747